CLINICAL TRIAL: NCT06250257
Title: Effect of Bromocriptine in Dilated Cardiomyopathy in Women of Reproductive Age: A Hospital-Based Randomized Open Label Placebo-controlled Clinical Trial
Brief Title: Bromocriptine in Dilated Cardiomyopathy Among Women of Reproductive Age
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jimma University (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Kedir Negesso Tukeni, Principal Investigator, Jimma University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JUIH/IRB/690/23
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Dilated Cardiomyopathy
Keywords: dilated cardiomyopathy; left ventricular function; ejection fraction; prolactin; bromocriptine; cardiac biomarkers; quality of life; Exercise capacity; 6-minute walk test; Standard stair climbing test
MeSH Terms: conditions — Cardiomyopathy, Dilated | interventions — Bromocriptine

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator): This group of study participants are expected to receive placebo (sucrose pills to be used) plus standard Guideline-directed medical therapy (GDMT).
  Interventions: Drug: Bromocriptine mesylate plus standard GDMT
- Treatment group (Experimental): This group of study participants are expected to receive oral daily bromocriptine 2.5 mg for 8 weeks plus standard Guideline-directed medical therapy (GDMT).
  Interventions: Drug: Bromocriptine mesylate plus standard GDMT

INTERVENTIONS:
Drug: Bromocriptine mesylate plus standard GDMT — The treatment group will receive bromocriptine 2.5mg PO daily for 8 weeks together with standard GDMT which include similar patterns of BBs, ACEI/ARBs, MRAs and SGLT2 inhibitors.

SUMMARY:
Dilated cardiomyopathy (DCM) is a condition associated with left and /or right ventricular (LV) dilatation and systolic dysfunction without coronary artery disease or abnormal loading circumstances proportionate to the severity of LV impairment. It is one of the leading causes of heart failure in younger adults. About 35% of patients have genetic mutations affecting cytoskeletal, sarcomere, and nuclear envelope proteins while others are idiopathic and possibly complications of myocarditis. Recently, in patients with peripartum cardiomyopathy (PPCM)-a subtype of dilated cardiomyopathy, high levels of prolactin and its degradation by-products including a cleaved 16kDa N-terminal fragment have emerged as key factors in the pathophysiology. The 16kDa prolactin induces profound endothelial damage and subsequent cardiomyocyte dysfunction and hence heart failure. Bromocriptine has been studied as a potential treatment option and placebo-controlled studies have demonstrated its beneficial role in women with Peripartal cardiomyopathy (PPCM). However, prolactin level may also increase during menstrual cycles of reproductive-age women, which candidates the use of bromocriptine in women of all reproductive ages. The aim of this study is therefore to assess the potential effect of bromocriptine in dilated cardiomyopathy among women of reproductive age.

DETAILED DESCRIPTION:
Background:

Cardiovascular diseases (CVDs) are the leading cause of death globally. An estimated 17.9 million people died from CVDs in 2017, representing 32% of all global deaths. Over three quarters of the CVD deaths take place in low- and middle-income countries. In 2022, CVDs account for almost 12% of the total burden of disease ranking third behind cancer and musculoskeletal conditions(1). A systematic review conducted in Ethiopia found that the prevalence of CVD ranges from 7.2 to 24% (2,3). Recently, the pooled prevalence of cardiovascular disease (CVD) was 5% (95% CI: 3-8%) with higher prevalence in the population who visits hospitals, 8% (95% CI: 4-12%) compared to the general population, 2% (95% CI: 1-5%) (3).

Dilated cardiomyopathy (DCM) is a condition associated with Left and or right ventricular (LV) dilatation and systolic dysfunction without coronary artery disease or abnormal loading circumstances proportionate to the severity of LV impairment (4-6). It is one of the leading causes of heart failure in younger adults, often requiring cardiac transplantation (7,8), and it is caused by various factors, including myocarditis, alcohol, drug, and metabolic disturbances (7,9). Hormonal factors including prolactin have recently been implicated to play a role in the development of DCM in women (10,11). About 35% of patients have genetic mutations affecting cytoskeletal, sarcomere, and nuclear envelope proteins while others are mainly idiopathic, including possibly complications of myocarditis (10-12). The prognosis depends on the severity and heart remodeling, with the worst outcomes in patients with low ejection fractions or severe diastolic dysfunction. DCM appears more common in men, than in women (12,13). However, a recent systematic review in Ethiopia indicates that there is no significant difference in the overall prevalence of CVD between males and females (3).

Despite many progresses made in the past decades in the development of novel pharmacological treatments for HF, proper management of HF is still challenging and there remains a substantial unmet need in heart failure. In recent years, a number of contributory mechanisms have been recognized to initiate and propagate cardiomyopathy (11-13). Prolactin has been found to be elevated in some cases of cardiomyopathy specially in the cases of peripartal cardiomyopathy (10,11), and may contribute to the development and progression of the condition. In patients with peripartum cardiomyopathy (PPCM), high levels of the hormone prolactin and the production of a cleaved 16kDa N-terminal fragment of prolactin have emerged as potential key factors in the pathophysiology of PPCM. The 16kDa prolactin induces profound endothelial damage and subsequent cardiomyocyte dysfunction and full-length prolactin promotes inflammation in PPCM (11-14).

Bromocriptine, a dopamine agonist that is primarily used to treat conditions such as Parkinson's disease, hyperprolactinemia, and acromegaly, has been investigated as a potential treatment option for Peripartal cardiomyopathy (PPCM), a form of DCM that occurs in the last month of pregnancy or up to five months postpartum (11,15). Clinical pilot studies showed the feasibility of bromocriptine in improving left ventricular (LV) recovery and clinical outcome (11,15-17). A recent multi-center randomized study comparing two different bromocriptine dosages (2.5 mg daily for one week vs. 5 mg daily for 2 weeks, followed by 2.5 mg daily for 6 weeks) in severe PPCM patients demonstrated an improved clinical outcome with high LV recovery rate at 6 months and with no mortality, no use of left ventricular assist device or heart transplantation (18,19).

Consequently, bromocriptine is recommended for the treatment of pregnancy-related cardiomyopathy (PPCM) due to a significant increase in prolactin levels in these group of patients. In such patients, the benefit of bromocriptine may be attributed to its ability to reduce prolactin levels. We hypothesize that, prolactin levels may also increase in women with DCM (15,19,20)of reproductive-age, and bromocriptine could also be a good candidate to use in women of all reproductive ages with DCM. Moreover, prolactin-independent cytoprotective effects of bromocriptine demonstrated in various organs including the heart may also support our hypothesis that bromocriptine may provide clinical benefit in all women with DCM (21-23).

Given the limited evidence to use of bromocriptine in DCM among women of reproductive age, further research is needed to fully understand whether or not bromocriptine improves clinical outcome compared to the standard treatment for heart failure in all or a subset of women. Therefore, this proposal aims to assess the potential benefit of bromocriptine in dilated cardiomyopathy among women of reproductive age. Thus, the study aims to provide a valuable information on the potential use of bromocriptine in women of reproductive age with DCM. If our hypothesis is confirmed, it may offer a good add-on treatment option that is also easily available for this population, and potentially improve treatment outcome and quality of life.

Problem statement

Heart failure (HF) is a progressively deteriorating medical condition that significantly reduces both patients' life expectancy and quality of life. Dilated cardiomyopathy (DCM) is one of the leading causes of heart failure in younger adults. Despite many progresses made in the past decades in the development of novel pharmacological treatments for HF, proper management of HF is still challenging and there remains a substantial unmet need in treating heart failure. Bromocriptine, an inhibiter of prolactin release by dopamine-D2-receptor, has been studied in the context of heart failure due to peripartal cardiomyopathy, and some studies have demonstrated its beneficial role in women with peripartum cardiomyopathy (PPCM) (15). As prolactin levels also increase in women of reproductive-age during menstrual cycle, bromocriptine could also be a good candidate to use in women of all reproductive ages and DCM.

Although reports show a beneficial role of bromocriptine in improving the left ventricular function in some patients with heart failure, the results may not be applicable to a wide range of populations and patients due to various sources of variation between populations (15) . Thus, it would be relevant to conduct a rigorous clinical trial to assess the efficacy and safety of this treatment option in diverse populations like Ethiopians in terms of etiologies of heart failure. It has been established that the same dose of a medication is associated with considerable heterogeneity in pharmacokinetics (PK) and pharmacodynamic (PD) efficacy and toxicity across human populations (16,17,21,23,24). This inter-individual difference in drug response can be explained by pharmacogenetic variations or other factors such as variations in patients' age and weight, co-morbidity, lifestyle, co-medication, renal and liver function, unfavorable drug-drug interactions and poor compliance of patients (17,24). The pharmacokinetics (PK) of bromocriptine in heart failure patients, the inter-individual variability in PK and clinical response and associated sources of variations have not been investigated before. Thus, this study is also designed to investigate the effectiveness of bromocriptine in terms of efficacy and safety as well as the blood levels and PK of bromocriptine among women of reproductive age with DCM in Ethiopia.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18 years to 50 years and
* ischemic or de novo dilated cardiomyopathy

Exclusion Criteria:

* Patients with severe comorbidities which may worsen their illness
* with hypertensive heart diseases
* Rheumatic valvular heart diseases
* Restrictive cardiomyopathy, constrictive cardiomyopathy, hypertrophic cardiomyopathy
* Congenital heart diseases
* Acute coronary syndrome
* Overt kidney failure (serum Creatinine ≥ 1.4mg/dl),
* Women who had history of peripartal cardiomyopathy, are pregnant or planning pregnancy during the study period or lactating
* Previous adverse reaction to the bromocriptine
* Patients not willing to participate in the study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — All women of reproductive age with diagnosis of dilated cardiomyopathy.
Enrollment: 112 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Left ventricular function improvement | at 3, 6 and 9 months
  Left ventricular function change measured in terms of ejection fraction and fractional shortening.
Improvement of cardiac biomarkers (N-terminal Pro BNP) | Measured at 3, 6 and 9 months
  Change in cardiac biomarkers measured as N-terminal Pro BNP.
Clinical improvement assessment tests | At recruitment, at 3,6, 9 and 12 months
  Exercise capacity improvement test with 6-minute walk test and stair climbing tests

SECONDARY OUTCOMES:
Change in hospitalization pattern | At 9 months and 1 year
  Change in hospitalization as compared with measurements before and after intervention
Functional class of heart failure Improvement | At 9 months and one year
  Change in NYHAF class as measured clinically and compared to the baseline status.
Improved quality of life | At 9 months and one year
  Change in quality of life as measured by Kansas City Cardiomyopathy Questionnaire (KCCQ-12) updated questionnaire, all KCCQ scores will be scaled from 0 to 100 and frequently summarized in 25-point ranges, where scores represent health status as follows: 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; and 75 to 100: good to excellent.

CONTACTS AND LOCATIONS:
Overall Officials: Kedir N Tukeni, MD, Principal Investigator — Jimma University; Haas A Nikolaus, MD, Cardiologist, Study Chair — Ludwig Maximillian university of Munich; Estner F Heidi, MD, cardiologist, Study Chair — Ludwig Maximillian university of Munich
Locations (1):
- Jimma Medical Center, Jimma, Oromiya, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
We will consider sharing the data after the completion of the study.
Supporting Information: CSR
Time Frame: We will share the data after the completion of the study till the study is published online.

REFERENCES:
- [Background] Vaideeswar P. Dilated Cardiomyopathy. In: Tropical Cardiovascular Pathology: Autopsy-Based Clinicopathological Cases. 2022
- [Background] Beg F, Wang R, Saeed Z, Devaraj S, Kamalesh M, Nakshatri H, et al. CIRCULATING FREE AND EXOSOMAL MICRORNAS AS BIOMARKERS OF SYSTEMIC RESPONSE TO HEART FAILURE. J Am Coll Cardiol. 2017;69(11).
- [Background] Eusuf D V., Thomas E. Pharmacokinetic variation. Vol. 23, Anaesthesia and Intensive Care Medicine. 2022.
- [Background] Sharma A, Klein AL. Diastolic Assessment: Application of the New ASE Guidelines. Vol. 11, Current Cardiovascular Imaging Reports. 2018.
- [Result] WHO CVD Risk Chart Working Group. World Health Organization cardiovascular disease risk charts: revised models to estimate risk in 21 global regions. Lancet Glob Health. 2019 Oct;7(10):e1332-e1345. doi: 10.1016/S2214-109X(19)30318-3. Epub 2019 Sep 2. PMID 31488387
- [Result] Misganaw A, Mariam DH, Ali A, Araya T. Epidemiology of major non-communicable diseases in Ethiopia: a systematic review. J Health Popul Nutr. 2014 Mar;32(1):1-13. PMID 24847587
- [Result] Angaw DA, Ali R, Tadele A, Shumet S. The prevalence of cardiovascular disease in Ethiopia: a systematic review and meta-analysis of institutional and community-based studies. BMC Cardiovasc Disord. 2021 Jan 18;21(1):37. doi: 10.1186/s12872-020-01828-z. PMID 33461482
- [Result] Peters S, Johnson R, Birch S, Zentner D, Hershberger RE, Fatkin D. Familial Dilated Cardiomyopathy. Heart Lung Circ. 2020 Apr;29(4):566-574. doi: 10.1016/j.hlc.2019.11.018. Epub 2019 Dec 17. PMID 31974027
- [Result] Eldemire R, Mestroni L, Taylor MRG. Genetics of Dilated Cardiomyopathy. Annu Rev Med. 2024 Jan 29;75:417-426. doi: 10.1146/annurev-med-052422-020535. Epub 2023 Oct 3. PMID 37788487
- [Result] Japp AG, Gulati A, Cook SA, Cowie MR, Prasad SK. The Diagnosis and Evaluation of Dilated Cardiomyopathy. J Am Coll Cardiol. 2016 Jun 28;67(25):2996-3010. doi: 10.1016/j.jacc.2016.03.590. PMID 27339497
- [Result] Pinto YM, Elliott PM, Arbustini E, Adler Y, Anastasakis A, Bohm M, Duboc D, Gimeno J, de Groote P, Imazio M, Heymans S, Klingel K, Komajda M, Limongelli G, Linhart A, Mogensen J, Moon J, Pieper PG, Seferovic PM, Schueler S, Zamorano JL, Caforio AL, Charron P. Proposal for a revised definition of dilated cardiomyopathy, hypokinetic non-dilated cardiomyopathy, and its implications for clinical practice: a position statement of the ESC working group on myocardial and pericardial diseases. Eur Heart J. 2016 Jun 14;37(23):1850-8. doi: 10.1093/eurheartj/ehv727. Epub 2016 Jan 19. PMID 26792875
- [Result] Reichart D, Magnussen C, Zeller T, Blankenberg S. Dilated cardiomyopathy: from epidemiologic to genetic phenotypes: A translational review of current literature. J Intern Med. 2019 Oct;286(4):362-372. doi: 10.1111/joim.12944. Epub 2019 Jul 29. PMID 31132311
- [Result] Pepperell RJ, Bright M, Smith MA. Serum prolactin levels in normal women and in women with disorders of menstruation. Med J Aust. 1977 Jan 22;1(4):85-9. doi: 10.5694/j.1326-5377.1977.tb130529.x. PMID 557719
- [Result] Hilfiker-Kleiner D, Kaminski K, Podewski E, Bonda T, Schaefer A, Sliwa K, Forster O, Quint A, Landmesser U, Doerries C, Luchtefeld M, Poli V, Schneider MD, Balligand JL, Desjardins F, Ansari A, Struman I, Nguyen NQ, Zschemisch NH, Klein G, Heusch G, Schulz R, Hilfiker A, Drexler H. A cathepsin D-cleaved 16 kDa form of prolactin mediates postpartum cardiomyopathy. Cell. 2007 Feb 9;128(3):589-600. doi: 10.1016/j.cell.2006.12.036. PMID 17289576
- [Result] Halkein J, Tabruyn SP, Ricke-Hoch M, Haghikia A, Nguyen NQ, Scherr M, Castermans K, Malvaux L, Lambert V, Thiry M, Sliwa K, Noel A, Martial JA, Hilfiker-Kleiner D, Struman I. MicroRNA-146a is a therapeutic target and biomarker for peripartum cardiomyopathy. J Clin Invest. 2013 May;123(5):2143-54. doi: 10.1172/JCI64365. Epub 2013 Apr 24. PMID 23619365
- [Result] Patten IS, Rana S, Shahul S, Rowe GC, Jang C, Liu L, Hacker MR, Rhee JS, Mitchell J, Mahmood F, Hess P, Farrell C, Koulisis N, Khankin EV, Burke SD, Tudorache I, Bauersachs J, del Monte F, Hilfiker-Kleiner D, Karumanchi SA, Arany Z. Cardiac angiogenic imbalance leads to peripartum cardiomyopathy. Nature. 2012 May 9;485(7398):333-8. doi: 10.1038/nature11040. PMID 22596155
- [Result] Sliwa K, Blauwet L, Tibazarwa K, Libhaber E, Smedema JP, Becker A, McMurray J, Yamac H, Labidi S, Struman I, Hilfiker-Kleiner D. Evaluation of bromocriptine in the treatment of acute severe peripartum cardiomyopathy: a proof-of-concept pilot study. Circulation. 2010 Apr 6;121(13):1465-73. doi: 10.1161/CIRCULATIONAHA.109.901496. Epub 2010 Mar 22. PMID 20308616
- [Result] Phillips KA, Veenstra DL, Oren E, Lee JK, Sadee W. Potential role of pharmacogenomics in reducing adverse drug reactions: a systematic review. JAMA. 2001 Nov 14;286(18):2270-9. doi: 10.1001/jama.286.18.2270. PMID 11710893
- [Result] Kumar A, Ravi R, Sivakumar RK, Chidambaram V, Majella MG, Sinha S, Adamo L, Lau ES, Al'Aref SJ, Asnani A, Sharma G, Mehta JL. Prolactin Inhibition in Peripartum Cardiomyopathy: Systematic Review and Meta-analysis. Curr Probl Cardiol. 2023 Feb;48(2):101461. doi: 10.1016/j.cpcardiol.2022.101461. Epub 2022 Oct 17. PMID 36261102
- [Result] Trongtorsak A, Kittipibul V, Mahabir S, Ibrahim M, Saint Croix GR, Hernandez GA, Chaparro S. Effects of bromocriptine in peripartum cardiomyopathy: a systematic review and meta-analysis. Heart Fail Rev. 2022 Mar;27(2):533-543. doi: 10.1007/s10741-021-10185-8. Epub 2021 Nov 1. PMID 34725781
- [Result] Samini M, Moezi L, Jabarizadeh N, Tavakolifar B, Shafaroodi H, Dehpour AR. Evidences for involvement of nitric oxide in the gastroprotective effect of bromocriptine and cyclosporin A on water immersion stress-induced gastric lesions. Pharmacol Res. 2002 Dec;46(6):519-23. doi: 10.1016/s1043661802002293. PMID 12457625
- [Result] Lim JH, Kim SS, Boo DH, No H, Kang BY, Kim EM, Hwang O, Choi HJ. Protective effect of bromocriptine against BH4-induced Cath.a cell death involving up-regulation of antioxidant enzymes. Neurosci Lett. 2009 Feb 27;451(3):185-9. doi: 10.1016/j.neulet.2008.12.056. Epub 2009 Jan 6. PMID 19146917
- [Result] Lim JH, Kim KM, Kim SW, Hwang O, Choi HJ. Bromocriptine activates NQO1 via Nrf2-PI3K/Akt signaling: novel cytoprotective mechanism against oxidative damage. Pharmacol Res. 2008 May;57(5):325-31. doi: 10.1016/j.phrs.2008.03.004. Epub 2008 Mar 22. PMID 18455424
- [Result] Gopalakrishnan P, Biederman R. Impact of the 2016 ASE/EACVI Guidelines on diastolic function reporting in routine clinical practice. Echocardiography. 2020 Apr;37(4):546-553. doi: 10.1111/echo.14645. Epub 2020 Apr 16. PMID 32298005
- [Result] Clancy DJ, Scully T, Slama M, Huang S, McLean AS, Orde SR. Application of updated guidelines on diastolic dysfunction in patients with severe sepsis and septic shock. Ann Intensive Care. 2017 Dec 19;7(1):121. doi: 10.1186/s13613-017-0342-x. PMID 29260409
- [Result] Lear SA, Brozic A, Myers JN, Ignaszewski A. Exercise stress testing. An overview of current guidelines. Sports Med. 1999 May;27(5):285-312. doi: 10.2165/00007256-199927050-00002. PMID 10368877
- [Result] Farrell MB. The Importance of Measurement for Quality Improvement: Submaximal Cardiac Stress Testing. J Nucl Med Technol. 2020 Jun;48(2):122-125. doi: 10.2967/jnmt.120.244525. Epub 2020 Apr 10. PMID 32277062
- [Result] Sullivan KM, Dean A, Soe MM. OpenEpi: a web-based epidemiologic and statistical calculator for public health. Public Health Rep. 2009 May-Jun;124(3):471-4. doi: 10.1177/003335490912400320. No abstract available. PMID 19445426
- Available data/document: Individual Participant Data Set — https://kf.kobotoolbox.org/#/forms/aSWyWhEb2TmCqshx54qTW7